CLINICAL TRIAL: NCT00814125
Title: A Randomised, Double Blind Trial to Assess the Incidence of Endometrial Changes With Arimidex Alone, Nolvadex Alone, or Arimidex and Nolvadex in Combination, When Used as Adjuvant Treatment for Breast Cancer in Postmenopausal Women
Brief Title: ATAC - Endometrial Sub-Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Francisco Sapunar, Medical Science Director, Arimidex and Faslodex, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1033IC/0029; D5392C06736
Record Dates: First submitted 2008-11-03; First posted 2008-12-24 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
Keywords: Endometrial; Endometrial histological findings
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Arimidex 1mg + Nolvadex placebo
  Interventions: Drug: Anastrozole (Arimidex); Drug: Nolvadex placebo
- 2 (Active Comparator): Arimidex placebo + Nolvadex 20mg
  Interventions: Drug: Tamoxifen (Nolvadex); Drug: Arimidex placebo
- 3 (Active Comparator): Arimidex 1mg + Nolvadex 20mg
  Interventions: Drug: Anastrozole (Arimidex); Drug: Tamoxifen (Nolvadex)

INTERVENTIONS:
Drug: Anastrozole (Arimidex) — 1mg, orally, once daily
  Other Names: Arimidex
  Arms: 1; 3
Drug: Tamoxifen (Nolvadex) — 20mg, orally, once daily
  Other Names: Nolvadex
  Arms: 2; 3
Drug: Nolvadex placebo
  Arms: 1
Drug: Arimidex placebo
  Arms: 2

SUMMARY:
To compare the difference between the ARIMIDEX group and the tamoxifen group in the incidence of abnormal endometrial histological findings arising after treatment has commenced.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for entry into the main ATAC trial (1033IL/0029)
* Not received any previous tamoxifen, for whatever reason
* Not undergone a hysterectomy and do not have a hysterectomy planned within the next 6 years
* No previous endometrial ablation

Exclusion Criteria:

* Excluded from entry into the main ATAC trial (1033IL/0029). As detailed in Section 4.4 of the main ATAC trial (1033IL/0029)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 1997-06; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Withdrawl
Death